CLINICAL TRIAL: NCT03420677
Title: Enhancement of Sleep Slow Wave Activity Using Wearable Auditory Stimulation Devices and Its Consequences on Daytime Functioning: a Randomized, Counter-balanced Crossover Study
Brief Title: Enhancement of Sleep With Wearables
Acronym: WESA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: WESA_2017-01436
Record Dates: First submitted 2017-12-04; First posted 2018-02-05 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Sleep

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application of tones (Active Comparator): During non-rapid eye movement (NREM) sleep short tones will be played
  Interventions: Device: Application of tones
- No application of tones (Sham Comparator): During NREM sleep no short tones will be played
  Interventions: Device: No application of tones

INTERVENTIONS:
Device: Application of tones — During NREM sleep, tones (max. 60 dB) will be played using a portable, safe, in-home device. This device records biosignals (e.g. brain activity) and precisely times the tones during NREM sleep. It was developed and produced by the ETH Zurich and approved for use in this study by Swissmedic
  Arms: Application of tones
Device: No application of tones — This is the sham-control intervention; The device will only record biosignals but will not play tones.
  Arms: No application of tones

SUMMARY:
Sleep, specifically deep sleep, plays a central role in healthy brain function, cardio-vascular processes, mood and quality of life. Auditory stimulation during one night of sleep has previously been shown to improve deep sleep and along with memory formation in both young and older adults. Yet, it remains unclear whether long-term auditory stimulation considerably improves sleep quality over longer time periods and how it affects daytime functioning such as cognition, mood, quality of life and peripheral functions (e.g. cardio-vascular). Due to the importance of deep sleep for brain and body and the presence of many conditions that involve reduced deep sleep (e.g. ageing) assessing the beneficial impact of long-term sleep enhancement and its consequences is of central interest.This study will assess the effect of auditory stimulation over two weeks (interleaved with a two weeks washout period) in a cohort of healthy young and older adults using portable recording and stimulation devices.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* For women: Hormonal contraception, if menstrual cycle is still present or has been present less than a year ago
* Good general health status
* Stable home situation (e.g. long-term place to live) that allows for reliable application of intervention for the duration of the study
* Male and Female subjects 18-35 years of age or 60-84 years of age
* German speaking

Exclusion Criteria:

* Women who are pregnant or breast feeding,
* Known or suspected non-compliance, drug or alcohol abuse,
* Intake of sleep altering medication
* Inability to follow the procedures of the study, e.g. due to language problems, cognitive deficits
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Presence or history of diagnosed psychiatric/neurologic disorder/lesion of the central nervous system (CNS),
* Diagnosed internal disease,
* Presence of sleep disorders,
* Shift-work (work during the night) or situations that require several awakenings during the night (e.g. newborn)
* Travelling more than 2 time zones in the last month before intervention starts or during intervention (study start will be shifted accordingly)
* Hearing disability/ hearing aid
* Skin disorders/problems in face region that will worsen with /not allow adhesive electrode application
* Nicotine/Cannabis use
* High caffeine consumption (> 5 servings/day; including coffee, energy drink)

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Sleep quality | From baseline period to study completion, assessed up to 2 months
  Objective information about sleep macro- and microstructure will be assessed including measures like sleep architecture, amount of slow wave activity (SWA), amount of spindles, awakenings during sleep, and sleep fragmentation. In addition, subjective sleep quality will be obtained by questionnaires every morning over the intervention period. These measures will show whether auditory stimulation enhanced overall sleep quality compared to sham.

SECONDARY OUTCOMES:
Daily functioning - Mood | From the beginning of the first intervention period until the end of the second intervention period, assessed within a time period up to 6 weeks
  Mood will be digitally assessed using a daily mood scale over the intervention period
Daily functioning - Quality of life | From the beginning of the first intervention period until the end of the second intervention period, assessed within a time period up to 6 weeks
  Quality of life will be assessed using a World Health Organization (WHO) quality of life assessment before and after each intervention period
Daily functioning - Vigilance | From the beginning of the first intervention period until the end of the second intervention period, assessed within a time period up to 6 weeks
  Vigilance will be assessed using a digital psychomotor vigilance task, assessed daily over the intervention period
Daily functioning - Cognition | From the beginning of the first intervention period until the end of the second intervention period, assessed within a time period up to 6 weeks
  Cognition will be assessed using a digital test battery before and after each intervention
Physiological parameters - Cardiovascular | From baseline period to study completion, assessed up to 2 months
  R-R interval based assessments will be obtained using wearable monitors
Physiological parameters - Physical activity | Through study completion, approximately 2 months
  Physical activity levels will be obtained using wearable monitors

OTHER OUTCOMES:
Device usability | From the first home visit until the end of the second intervention period, assessed within a time period up to 2 months
  Questionnaires will be used to track specific information about the portable intervention device including information about its usability, discomfort and blinding to the condition
Diary | Through study completion, approximately 2 months
  Information about daily habits will be digitally assessed
Incidence of Intervention-related Adverse Events [Safety and Tolerability] | Through study completion, approximately 2 months
  Any adverse or serious adverse events during the study period will be assessed
Chronotype | Before start of intervention period (single-time assessment during one initial 1-day visit)
  Assessment of circadian type
Handedness | Before start of intervention period (single-time assessment during one initial 1-day visit)
  Assessment of handedness
Menstrual cycle | Before start of intervention period (single-time assessment during one initial 1-day visit)
  Assessment of menstrual cycle information in woman
Height | Before start of intervention period (single-time assessment during one initial 1-day visit)
  Assessment of height
Hip-to-waist ratio | Before start of intervention period (single-time assessment during one initial 1-day visit)
  Assessment of hip and waist circumference
Blood pressure | Through study completion, approximately 2 months
  Assessment of blood pressure
Weight | Before start of intervention period (single-time assessment during one initial 1-day visit)
  Assessment of weight

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Federal Institute of Technology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Lustenberger C, Ferster ML, Huwiler S, Brogli L, Werth E, Huber R, Karlen W. Auditory deep sleep stimulation in older adults at home: a randomized crossover trial. Commun Med (Lond). 2022 Apr 4;2:30. doi: 10.1038/s43856-022-00096-6. eCollection 2022. PMID 35603302